CLINICAL TRIAL: NCT07233746
Title: Comparison of the Effects of Quadroiliac Plane Block Versus Suprainguinal Fascia Iliaca Compartment Block on Postoperative Pain in Hip Surgery
Brief Title: Comparison of QIPB and SIFICB in Hip Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Associate Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2025-07/23
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain; Hip Surgery
Keywords: postoperative pain; hip surgery; regional anesthesia; quadroiliac plane block; suprainguinal fascia iliaca compartment block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadro-İliac Plane Block(QİPB) (Active Comparator): For this group, after the surgical procedure is completed, the patient will be placed in a lateral position with the operated side facing up, and a QIPB will be performed. With the patient in the lateral position, the spinous process of the L3 vertebra will first be imaged with an ultrasound probe positioned transversely in the midline. Then, by slightly shifting the probe laterally, the transverse process of the vertebra will be visualized within the erector spinae muscle. The probe will then be rotated in the sagittal plane and advanced caudally about 1 cm, visualizing the crista iliaca. On the cranial side of the crista iliaca, the erector spinae muscle, quadratus lumborum, and psoas major muscles will be visualized sequentially. With the needle direction cranial to caudal, the crista iliaca will be gently touched, and the needle will be positioned between the erector spinae and the quadratus lumborum muscle. After injecting 40 ml of 0.25% bupivacaine, the needle will be injected.
  Interventions: Procedure: Quadro-İliac Plane Block(QİPB)
- Suprainguinal Fascia Iliaca Compartiment Block (SIFICB) (Active Comparator): Probe Placement: A high-frequency linear ultrasound probe is placed in a sagittal orientation over the Anterior Superior Iliac Spine (ASIS) and then moved medially.
  Anatomical Landmark: The key visual target on the ultrasound screen is the "bowtie" sign, which is formed by the junction of the sartorius and internal oblique muscles over the iliacus muscle.Injection Point: The target for injection is the potential space located directly beneath the fascia iliaca (seen as a bright, hyperechoic line) and superficial to the iliacus muscle.Needle Insertion: The block needle is advanced using an "in-plane" technique (parallel to the probe's long axis), typically from a caudal-to-cranial direction (from bottom to top).Injection: After confirming correct needle tip placement with hydrodissection (visualizing fluid separating the fascia from the muscle), 30-40 mL of local anesthetic is slowly injected. The spread of the anesthetic proximally (upward) beneath the fascia is monitored in real-time
  Interventions: Procedure: Suprainguinal Fascia Iliaca Compartiment Block

INTERVENTIONS:
Procedure: Quadro-İliac Plane Block(QİPB) — 40 mL of 0.25% bupivacaine
  Arms: Quadro-İliac Plane Block(QİPB)
Procedure: Suprainguinal Fascia Iliaca Compartiment Block — 30 mL of 0.25% bupivacaine
  Arms: Suprainguinal Fascia Iliaca Compartiment Block (SIFICB)

SUMMARY:
The aim is to compare the postoperative analgesic effects of Quadroiliac Plane Block (QIPB) and Suprainguinal Fascia Iliaca Compartment Block (SIFICB) in patients undergoing hip surgery.

DETAILED DESCRIPTION:
Patients were divided into two randomized groups: Group 1 (QIPB group, n=30) and Group 2 (SIFICB group, n=30). All patients will receive the same standard general anesthesia per hospital protocol. All blocks will be applied with the same ultrasonography and block equipment, and by the same physician. After the anesthesia induction, patients in Group 1 will receive Quadroiliac Plane Block (QIPB) with 40 mL of 0.25% bupivacaine. Patients in Group 2 will receive Suprainguinal Fascia Iliaca Compartment Block (SIFICB) with 30 mL of 0.25% bupivacaine. All patients will receive Paracetamol 1gr and Dexketoprofen 50mg intravenous (IV) 10 minutes prior to skin closure. Routine analgesic procedure consisting of 3x400mg Ibuprofen will be followed postoperatively for 24 hours. Numeric Rating Scale (NRS) will be used to assess postoperative pain on 1st, 6th, 12th, 18th and 24th hours after the surgery. Tramadol 1mg/kg IV will be administered as a rescue analgesic for all patients if NRS score is higher than 4. Total Tramadol consumption will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age who underwent percutaneous nephrolithotomy under general anesthesia and were I-II-III according to the American Society of Anesthesiologists (ASA) risk classification were included in the study.

Exclusion Criteria:

* patients who did not give consent,

  * patients with coagulopathy,
  * patients with signs of infection at the block application site,
  * patients using anticoagulants,
  * patients with known allergies to any of the study drugs,
  * patients with unstable hemodynamics,
  * patients who could not cooperate during postoperative pain assessment
  * patients who wanted to withdraw from the study,
  * patients with alcohol and drug addiction,
  * patients with musculoskeletal abnormalitie

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) Scores | Postoperative 24 hours
  Numerical rating scale is used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Total tramadol consumption | Postoperative 24 hours
  Postoperative total analgesic need was recorded as "milligram" in unit.

CONTACTS AND LOCATIONS:
Overall Officials: OĞUZ GÜNDOĞDU, Principal Investigator — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation; MAHMUT K DEMİRCİ, Study Chair — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation
Locations (1):
- Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation, Sivas, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No